CLINICAL TRIAL: NCT04154709
Title: CTA101 UCAR-T Cell Injection for Treatment of Relapsed or Refractory CD19+ B-cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kai Lin Xu; Jun Nian Zheng (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Kai Lin Xu; Jun Nian Zheng, President, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2019-KL135-02
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTA101 (Experimental): Dose escalation follows the accelerated titration and the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Biological: CTA101

INTERVENTIONS:
Biological: CTA101 — Universal CD19-directed CAR-T cells by a single infusion intravenously will be given in escalating doses.

SUMMARY:
This study aims to evaluate the safety and feasibility of CTA101 in treating patients with relapsed or refractory CD19+ B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
This study is indicated for r/r CD19+ B-ALL, the selection of dose levels and the number of subjects are based on clinical trial of similar foreign product, whose primary objective was to explore the safety, main consideration was dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 3-70 years old;
2. Histologically confirmed diagnosis of CD19+ B-ALL per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (2016.v1);
3. Relapsed or refractory CD19+ B-ALL (meeting one of the following conditions):

   1. CR not achieved after standardized chemotherapy;
   2. CR achieved following the first induction, but CR duration is ≤ 12 months;
   3. Ineffectively after first or multiple remedial treatments;
   4. 2 or more recurrences;
4. The number of primordial cells (lymphoblast and prolymphocyte) in bone marrow is﹥5%;
5. Philadelphia-chromosome-negative (Ph-) patients; or Philadelphia-chromosome-positive (Ph+) patients who cannot tolerate TKI treatments or do not respond to 2 TKI treatments;
6. Serum albumin ≥ 30g/L, total bilirubin ≤ 25.7umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8umol/L, platelet count ≥ 50*10^9/L;
7. Echocardiogram (ECHO) shows left ventricular ejection fraction (LVEF) ≥ 50%;
8. No active infection in the lungs, blood oxygen saturation in indoor air is ≥ 92%;
9. Latest treatment (radiotherapy, chemotherapy, monoclonal antibody therapy or other treatment) must have been completed at least 2 weeks prior to screening;
10. Estimated survival time ≥ 3 months;
11. ECOG performance status 0 to 1;
12. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

1. History of hypersensitivity to any component of cell product;
2. Prior treatment with any CAR T cell product or other genetically-modified T cell therapies;
3. Patients with extramedullary lesions;
4. Confirmed diagnosis of lymphoblastic crisis of chronic myeloid leukemia, Burkitt's leukemia/ lymphoma per WHO Classification Criteria;
5. Patients with hereditary syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome;
6. Patients with New York Heart Associate (NYHA) Class III/IV cardiac insufficiency;
7. Myocardial infarction, cardioangioplasty or stenting, unstable angina pectoris, or other severe cardiac diseases within 12 months of enrollment;
8. Severe primary or secondary hypertension of grade 3 or above (WHO Hypertension Guidelines, 1999);
9. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
10. Central nervous system leukemia (CNS2 or CNS3), resistant to intrathecal injecting of chemotherapeutic drugs, and/or undergoing skull and/or spine radiotherapy; patients with history of CNS but effectively controlled to allow enrollment;
11. Prior treatment with TKIs (Ph+ ALL) 1 week prior to enrollment;
12. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis), or currently receiving antibiotic therapy by intravenous infusion, or have received antibiotic treatment by intravenous infusion within 1 week before cell infusion. However, prophylactic antibiotic, antiviral and antifungal treatments are allowed;
13. Indwelling catheters in vivo (e.g. percutaneous nephrostomy, Foley catheter, bile duct catheter, or pleural/peritoneal/pericardial catheter). Ommaya storage, dedicated central venous access catheters such as Port-a-Cath or Hickman catheters are allowed;
14. History of other primary cancer, except for the following conditions:

    1. Cured non-melanoma after resection, such as basal cell carcinoma of the skin;
    2. Cervical cancer in situ, localized prostate cancer, ductal cancer in situ with disease-free survival ≥ 2 years after adequate treatment;
15. Patients with autoimmune diseases requiring treatment, patients with immunodeficiency or requiring immunosuppressive therapy;
16. Patients with graft-versus-host disease (GVHD);
17. If HBsAg positive at screening, HBV DNA copy number detected by PCR in patients with active hepatitis B > 1000 (if HBV DNA copy number≤1000, routine antiviral therapy is required after enrollment), as well as CMV, hepatitis C, syphilis and HIV infection;
18. Concurrent therapy with systemic steroids within 1 week prior to screening, except for the patients recently or currently receiving inhaled steroids;
19. Women pregnant or lactating, with a pregnancy plan within 6 months, fertile but unable to take medically acceptable contraception measures.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | Baseline up to 28 days after T cell infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
MRD negative overall response rate (MRD- ORR) | 3 months
  Assessment of MRD negative overall response rate (MRD- ORR) at 3 months of treatment
Overall response rate (ORR) | Month 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi ) at Month 6, 12, 18 and 24
Event-free survival (EFS) | Month 6, 12, 18 and 24
  Assessment of EFS at Month 6, 12, 18 and 24
Overall survival (OS) | Month 6, 12, 18 and 24
  Assessment of OS at Month 6, 12, 18 and 24

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of Xuzhou medical college, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No